CLINICAL TRIAL: NCT03081559
Title: Improving Engagement in HIV Care for High-risk Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH106373 (NIH)
Record Dates: First submitted 2017-03-06; First posted 2017-03-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: HIV/AIDS; Adherence, Medication
Keywords: transgender; women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Healthy Divas intervention
  Interventions: Behavioral: Healthy Divas
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Healthy Divas — Peer-based counseling to improve medication adherence and engagement in care
  Arms: Intervention

SUMMARY:
Transgender women (assigned 'male' at birth but who do not identify as male) are disproportionately impacted by HIV and have culturally unique barriers and facilitators to engagement in HIV care. Transgender women living with HIV (TWH) are less likely than others to take antiretroviral therapy (ART), and those who initiate ART have lower rates of ART adherence, lower self-efficacy for integrating ART into daily routines, and report fewer positive interactions with health care providers than non-transgender adults. As a result, TWH have an almost three-fold higher viral load than non-transgender adults in San Francisco; in Los Angeles, TWH are less likely to be virally suppressed than any other behavioral risk group. In formative work, the investigators have identified culturally-specific and modifiable barriers to HIV treatment engagement among TWH, including prioritization of transition-related health care (i.e. hormone therapy) at the expense of HIV treatment, avoidance of HIV care settings due to past negative health care experiences, misinformation about ART including potential drug interactions with hormones, intensified HIV stigma, low levels of social support, and poor coping skills. There are both individual and public health consequences to poor engagement in care among TWH stemming from high transmission risk factors, including substance abuse, high numbers of sex partners, engagement in sex work, and high rates of mental illness. These findings strongly suggest that TWH face unique challenges to engaging in and adhering to HIV treatment, and that the public health consequences for poor engagement in this population are of grave concern. Interventions to mitigate these barriers to engagement in care are critical in efforts to alter the pattern of HIV-related disparities that lead to disproportionately poor health outcomes for this highly vulnerable and marginalized population. The investigators are conducting a randomized controlled trial of a theory-driven, population-specific, piloted intervention to improve engagement in care for TWH. Grounded in the investigators' Models of Gender Affirmation and Health Care Empowerment, the proposed research is the first to systematically intervene on complex barriers to optimal engagement in HIV care for TWH. The investigators have developed and piloted the Healthy Divas intervention to optimize engagement in HIV care for TWH at elevated risk for treatment failure and consequential morbidity, mortality, and transmission of HIV.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years old; and
2. Assigned male sex at birth but does not currently identify as male; and
3. English- or Spanish-speaking; and
4. HIV+ confirmed via antibody testing; and
5. Evidence of suboptimal engagement in HIV care, as indicated by one or more of the following:

   1. Not on ART; (b) If on ART, reporting less than perfect adherence on a validated adherence rating scale; or (c) Reporting no HIV primary care appointments in the prior 6 months.

Exclusion Criteria:

Evidence of severe cognitive impairment or active psychosis, as determined by the Project Director in consultation with the Principal Investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women
Enrollment: 278 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change in virologic control | Baseline, 3, 6, 9, 12 months
  As indicated by an undetectable HIV-1 level on the COBAS® AmpliPrep/COBAS® TaqMan® HIV test kit (Roche Molecular Systems, Inc.)

SECONDARY OUTCOMES:
Change in behavioral composite of engagement in HIV care | Baseline, 3, 6, 9, 12 months
  Composite measure which integrates current/past ART use, HIV appointments timeline followback , ART adherence (adherence rating and visual analog scale), and knowledge of current CD4 cell count.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Sevelius, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Friends Community Center, Los Angeles, California
  - Alliance Health Project, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sevelius J, Veras MASM, Gomez JL, Saggese G, Mocello AR, Bassichetto KC, Neilands TB, Lippman SA. Reducing intersectional stigma among transgender women in Brazil to promote uptake of HIV testing and PrEP: study protocol for a randomised controlled trial of Manas por Manas. BMJ Open. 2024 Jun 21;14(6):e076878. doi: 10.1136/bmjopen-2023-076878. PMID 38908840
- [Derived] Sevelius JM, Neilands TB, Reback CJ, Castro D, Dilworth SE, Kaplan RL, Johnson MO. An Intervention by and for Transgender Women Living With HIV: Study Protocol for a Two-Arm Randomized Controlled Trial Testing the Efficacy of "Healthy Divas" to Improve HIV Care Outcomes. Front Reprod Health. 2021 Oct 27;3:665723. doi: 10.3389/frph.2021.665723. eCollection 2021. PMID 36304034
- [Derived] Sevelius JM, Dilworth SE, Reback CJ, Chakravarty D, Castro D, Johnson MO, McCree B, Jackson A, Mata RP, Neilands TB. Randomized Controlled Trial of Healthy Divas: A Gender-Affirming, Peer-Delivered Intervention to Improve HIV Care Engagement Among Transgender Women Living With HIV. J Acquir Immune Defic Syndr. 2022 Aug 15;90(5):508-516. doi: 10.1097/QAI.0000000000003014. Epub 2022 Mar 5. PMID 35502891